CLINICAL TRIAL: NCT01665339
Title: Effect of Preload on Body Weight and Cardiovascular Risks
Brief Title: Preload, Weight Management, Risk of Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Principal Investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Effect of preload on weight; IUMS (Other: Isfahan University of Medical Sciences)
Record Dates: First submitted 2012-08-01; First posted 2012-08-15 (Estimated); Last update posted 2012-08-15 (Estimated); Status verified 2012-08

CONDITIONS: Body Weight
Keywords: preload; anthropometric measures; cardiovascular risk factors
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- preload (Experimental): subjects in preload group consumed salad, yogurt and water 15 minutes before the main meal.
  Interventions: Other: preload diet
- control (Experimental): subjects in control group consumed salad and yogurt with meal.
  Interventions: Other: control diet

INTERVENTIONS:
Other: preload diet — All participants were prescribed a calorie-restricted diet (-200 to -500 kcal/d). Calorie requirements of each subject were estimated based on resting energy expenditure (REE) by using Harris- Benedict equation and also considering the physical activity levels. The diets were constructed to provide similar proportions of carbohydrates (55% energy), protein (15% energy) and total fat (30% energy).
  Arms: preload
Other: control diet — All participants were prescribed a calorie-restricted diet (-200 to -500 kcal/d). Calorie requirements of each subject were estimated based on resting energy expenditure (REE) by using Harris- Benedict equation and also considering the physical activity levels. The diets were constructed to provide similar proportions of carbohydrates (55% energy), protein (15% energy) and total fat (30% energy).
  Arms: control

SUMMARY:
Investigators presumed that preload consumers will have more weight reduction and lower risk of cardiovascular disease

DETAILED DESCRIPTION:
To our knowledge, all previous studies evaluated the energy intake in a dietary meal after consuming a low-energy-dense preload while none assessed the sustainability of lower amount of energy intake and body weight changes in a long-term. On the other hand, the sustainability of lower energy intake in a long term might be affected by higher dietary diversity score due to considering preload in diets. Notably, increased diet variety is associated with higher overall dietary energy intake and weight gain.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25,
* older than 18 years

Exclusion Criteria:

* poor dietary compliance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
the amount of weight reduction in two dietary groups | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Leila Azadbakht, PhD, Principal Investigator — Isfahan University of Medical Sciences